CLINICAL TRIAL: NCT06927570
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-20122 in Patients With Advanced Solid Tumors
Brief Title: A Study of HS-20122 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20122-101
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; HS-20122

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-20122 (Experimental): All subjects will receive HS-20122 in a continuous regimen in dose escalation stage or dose expansion stage
  Interventions: Drug: HS-20122

INTERVENTIONS:
Drug: HS-20122 — Intravenous (IV) administration of HS-20122 ; Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and confirmed disease progression.

SUMMARY:
This is a first-in-human (FIH) Phase I, multi-center, open-label, study of HS-20122, in patients with advanced solid tumors. This study will evaluate the safety, tolerability, pharmacokinetics and efficacy of HS-20122 in advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years.
* Subjects with histologically or cytologically confirmed locally advanced or metastatic Solid Tumors
* Standard treatment is invalid, unavailable or intolerable.
* At least 1 target lesion according to RECIST 1.1.
* ECOG PS score: 0-1.
* Estimated Life expectancy> 12 weeks.
* Men or women should be using adequate contraceptive measures throughout the study.
* Women must have the evidence of non-childbearing potential.
* Signed and dated Informed Consent Form.

Exclusion Criteria:

* Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 with the exception of alopecia or neurotoxicity
* History of other primary malignancies.
* Inadequate bone marrow reserve or organ dysfunction.
* Evidence of cardiovascular risk.
* Subjects with severe or poorly controlled diabetes.
* Subjects with severe or poorly controlled hypertension.
* Subjects with clinically significant bleeding symptoms or obvious bleeding tendency within 1 month prior to the first dose.
* Subjects with severe arteriovenous thrombotic events within 3 months.
* Subjects with severe infection within 4 weeks prior to the first dose.
* Subjects who have received steroid therapy for more than 30 days .
* Presence of known active infectious diseases.
* Presence of clinically significant gastrointestinal dysfunction.
* Hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis ≥ Child-Pugh Grade B.
* Moderate to severe pulmonary diseases.
* Prior history of significant neurological or mental disorders.
* Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
* Hypersensitivity to any ingredient of HS-20122.
* Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
* Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments Any unresolved toxicities from prior therapy greater than Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0 with the exception of alopecia or neurotoxicity
* History of other primary malignancies.
* Inadequate bone marrow reserve or organ dysfunction.
* Evidence of cardiovascular risk.
* Subjects with severe or poorly controlled diabetes.
* Subjects with severe or poorly controlled hypertension.
* Subjects with clinically significant bleeding symptoms or obvious bleeding tendency within 1 month prior to the first dose.
* Subjects with severe arteriovenous thrombotic events within 3 months.
* Subjects with severe infection within 4 weeks prior to the first dose.
* Subjects who have received steroid therapy for more than 30 days .
* Presence of known active infectious diseases.
* Presence of clinically significant gastrointestinal dysfunction.
* Hepatic encephalopathy, hepatorenal syndrome, or liver cirrhosis ≥ Child-Pugh Grade B.
* Moderate to severe pulmonary diseases.
* Prior history of significant neurological or mental disorders.
* Women who are breastfeeding or pregnant or planned to be pregnant during the study period.
* Hypersensitivity to any ingredient of HS-20122.
* Unlikely to comply with study procedures, restrictions, and requirements in the opinion of the investigator
* Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) or the maximum applicable dose (MAD) | From time of first dose of HS-20122 to end of DLT period (approximately 21 days)
  To determine the MTD or MAD for further evaluation of intravenous administration of HS-20122 in subjects with advanced solid tumors

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From time of Informed Consent to 28 days post last dose of HS-20122
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
Incidence of dose-limiting toxicities (DLT) as defined in the protocol | From time of first dose of HS-20122 to end of DLT period (approximately 21 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Observed maximum drug concentration (Cmax) of HS-20122 (including antibody-drug conjugates, total antibody, and payload) | From the date of first dose until 30 days after the final dose
  The Cmax is the maximum observed drug concentration of HS-20122
Time to reach maximum observed drug concentration (Tmax) of HS-20122 (including antibody-drug conjugates, total antibody, and payload) | From the date of first dose until 30 days after the final dose.
  The Tmax is defined as time to reach maximum observed drug concentration of HS-20122.
Area under the curve from time Zero to end of dosing interval (AUC0-t) of HS-20122 (including antibody-drug conjugates, total antibody, and payload) | From the date of first dose to Cycle 4(each cycle is 28 days) pre-dose.
  The AUC0-t is defined as the area under the drug concentration-time curve during a dose interval time period(t)
Area under the curve from time Zero to end of dosing interval (AUC0-∞) of HS-20122 (including antibody-drug conjugates, total antibody, and payload) | From the date of first dose to Cycle 4(each cycle is 28 days) pre-dose
  The AUC0-∞ is defined as the area under the drug concentration-time curve from time 0 to infinity
Incidence of anti-HS-20122 antibody (ADA) | From the date of first dose until 30 days after the final dose.
  ADA incidence was defined as the percentage of participants whose ADA status were identified as positive.
Objective response rate (ORR) | up to 24 months
  ORR was defined as the percentage of participants who achieved a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR), assessed by investigators based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China